CLINICAL TRIAL: NCT00236587
Title: An Open Label, Long Term Trial of Risperidone Long Acting Microspheres in the Treatment of Patients Diagnosed With Schizophrenia
Brief Title: A Long Term Study of Long-acting Injectable Risperidone in the Treatment of Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003274
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Intramuscular injection; Antipsychotic agents; Long-acting risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to document the long term safety of a long-acting injectable formulation of risperidone in the treatment of patients with schizophrenia who have previously been treated with long-acting risperidone. Efficacy will also be evaluated.

DETAILED DESCRIPTION:
This is an open-label, long-term study of a flexible dose of a long-acting injectable formulation of risperidone (risperidone LAI) injected into the muscle at 2 week intervals for at least 12 months in patients diagnosed with schizophrenia. It is an extension of an open label study of patients with schizophrenia (RIS-USA-259) switching from treatment with an oral antipsychotic medication to long-acting injectable risperidone. Safety evaluations include incidence of adverse events, physical examinations, clinical laboratory tests (biochemistry, hematology, and urinalysis), electrocardiograms (ECGs), and Extrapyramidal Symptom Rating Scale (ESRS), a scale for assessing muscle tone, gait, and abnormal movements. Efficacy assessments include measurements using the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) and the Clinical Global Impression-Severity of Illness scale (CGI-S). Risperidone (25-50milligrams [mg]) injections, long-acting formulation, every 2 weeks for at least 1 year. Dosages may be increased (50 mgs maximum) or decreased at discretion of the investigator. Supplementary risperidone tablets (1mg) may be administered.

ELIGIBILITY:
Inclusion Criteria:

* Completion of RIS-USA-256 within 7 days

Exclusion Criteria:

* History of neuroleptic malignant syndrome, a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness
* Significant and untreated or unstable medical illness such as diabetes, hypertension, angina
* Serious illness of the liver, kidney, or significant disturbances of the cardiac, pulmonary, gastrointestinal, endocrine, neurological system
* Pregnant or nursing females, or those lacking adequate contraception
* Known hypersensitivity or unresponsiveness to risperidone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-11; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
To accumulate long-term safety data: incidence of adverse events and clinical evaluations (physical examination, Extrapyramidal Symptom Rating Scale [ESRS], laboratory tests, ECGs).

SECONDARY OUTCOMES:
To evaluate long-term efficacy: Positive and Negative Syndrome Scale for Schizophrenia and the Clinical Global Impression-Severity of Illness subscale (CGI-S) every 3 months, including last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A long term study of long-acting injectable risperidone in the treatment of patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=517&filename=CR003274_CSR.pdf